CLINICAL TRIAL: NCT05082415
Title: Real-world Evaluation of Brolucizumab for the Treatment of Neovascular (Wet) Age-related Macular Degeneration (AMD) (IRIS Study)
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CRTH258AUS15
Record Dates: First submitted 2021-10-05; First posted 2021-10-19 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2021-10

CONDITIONS: Age-related Macular Degeneration (AMD)
Keywords: Brolucizumab,; intravitreal injection,; neovascular age-related macular degeneration,; visual acuity
MeSH Terms: conditions — Macular Degeneration | interventions — brolucizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Brolucizumab: Participants received brolucizumab injection during the index period
  Interventions: Drug: Brolucizumab

INTERVENTIONS:
Drug: Brolucizumab — Participants received brolucizumab injection during the index period
  Other Names: BEOVU®

SUMMARY:
This study was a retrospective cohort study of patients to assess the early insights into real-world safety among wet AMD patients initiating brolucizumab. Evidence was generated to describe their patient characteristics and clinical outcomes. The study was conducted using the IRIS Registry.

DETAILED DESCRIPTION:
IRIS Registry EHR data from patients with wet AMD who initiated brolucizumab were analyzed in this study.

Identification period of the index date (index period): The patients fulfilling the selection criteria was identified

* Index date: Defined as the date of the earliest brolucizumab injection
* Study Period: The period from the first patient eye exposure to brolucizumab to the last follow-up recorded
* Pre-index period: The period 36 months prior to the index date. Data within 36 months prior to the index date will be used to assess baseline characteristics.
* Post-index period: The period 180 days after the index date

ELIGIBILITY:
Inclusion Criteria:

1. ≥1 Healthcare Common Procedure Coding System (HCPCS) code (J code) or EMR note for treatment with brolucizumab during the index period (date of earliest code or EMR note = index date)
2. ≥18 years old on the index date
3. ≥1 Current Procedural Terminology (CPT) code for intravitreal administration on the index date
4. ≥1 International Classification of Diseases, Clinical Modification-9/10 (ICD-9/10) code for wet AMD in the 36 months prior to or on the index date

   o Note: Off-label use of brolucizumab is not expected given payer access restrictions in the US.
5. ≥1 follow-up visit after the index date
6. ≥1 VA assessment on the index date or within 90 days prior to the index date

Exclusion Criteria:

1. Use of brolucizumab prior to 10/8/2019 (e.g. clinical trials)
2. Unknown laterality of the index eye on the index date

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with wet AMD who initiated brolucizumab were analyzed in this study.
Sampling Method: Non-Probability Sample
Enrollment: 9456 (Actual)
Dates: Start 2020-06-03 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
Number of patient eyes with an Intraocular Inflammation (IOI) event during the first 6 months | Up to 6 months post brolucizumab injection
  To assess IOI events observed after starting treatment with brolucizumab

SECONDARY OUTCOMES:
Age | At the brolucizumab index date defined as the date of first brolucizumab injection
  Age information was reported
Gender information | At the brolucizumab index date defined as the date of first brolucizumab injection
  Gender information was reported
Number of patients at various Patient Region | At the brolucizumab index date defined as the date of first brolucizumab injection
  Patient regions: Northeast, Midwest, South, West, Unknown
Number of patients with Insurance type | At the brolucizumab index date defined as the date of first brolucizumab injection
  Insurance type: Medicare, Medicare Advantage, Medicaid, Commercial, Government, Military, No Insurance, Miscellaneous, Unknown
Number of patients with Laterality of wet Age-related macular degeneration (AMD) | At the brolucizumab index date defined as the date of first brolucizumab injection
  Laterality of wet AMD: Unilateral, Bilateral
Race/Ethnicity of the participants (patient level and eye level) | At the brolucizumab index date defined as the date of first brolucizumab injection
  Caucasian, Black or African American, Asian, Other, Unknown
Number of eyes with the concurrent eye disease | Within 180 days prior to the index date (inclusive of the index date) ( index date defined as the date of first brolucizumab injection)
  Types of concurrent eye diseases: ▪ Cataracts
  * Posterior vitreous detachment
  * Puckering of macula
  * Macular hole
  * Vitreomacular traction
  * Glaucoma
  * Amblyopia
  * Papillitis
  * Ischemic optic atrophy
  * Diabetic retinopathy
  * Diabetic macular edema
  * Hypertensive retinopathy
  * Pathologic myopia
  * RAO
  * RO
  * RV
  * Vitritis
  * Endophthalmitis
  * Uveitis
  * Choroidal neovascularization (due to causes other than AMD, if possible, to determine)
  * IOI
Number of patient eyes with cataract status | 36-month period prior to the index date (inclusive of the index date) ( index date defined as the date of first brolucizumab injection)
  Types: phakic, pseudophakic, aphakic
Number of patient eyes with Concomitant ocular medications | 36-month period prior to the index date (inclusive of the index date) ( index date defined as the date of first brolucizumab injection)
  Types:
  * Corticosteroids
  * Prednisone
  * Prednisolone acetate
  * Difluprednate
  * Biologics
  * Cyclosporine
  * Methotrexate
  * Ganciclovir
  * Acyclovir
  * Trifluridine
  * Rituxan
Number of patient eyes with the history of ocular inflammation | 36-month period prior to the index date (inclusive of the index date) ( index date defined as the date of first brolucizumab injection)
  The following categories were reported:
  * No history of inflammation
  * History of any ocular inflammation
  * History of severe ocular inflammation
  * History of anterior inflammation
  * History of posterior inflammation
  * History of IOI or endophthalmitis due to infections and other underlying disease (separate category)
Number of patient eyes with prior Intraocular Inflammation (IOI) and/or prior Retinal vascular occlusion (RO) | 12 months prior to the index date ( index date defined as the date of first brolucizumab injection)
  Included history of ocular inflammation or occlusion
Number of patient eyes with the Provider specialty | At the brolucizumab index date defined as the date of first brolucizumab injection
  The following types were included:
  Retina specialist, General ophthalmologist, Non-retina specialist, unknown
Number of patient eyes with the previous ocular surgeries or procedures | 6 months prior to the index date ( index date defined as the date of first brolucizumab injection)
  The following categories were included:
  * Laser therapy
  * Laser coagulation
  * Photodynamic therapy
  * IOP lowering surgeries (lasers, glaucoma filtering, non-filtering glaucoma)
  * Cataract surgery
  * Iridotomy
  * Intraocular or refractive surgery (almost all IOP & cataract surgeries)
  * Previous penetrating keratoplasty, vitrectomy, or ocular radiation
  * Previous panretinal photocoagulation
  * Previous submacular surgery, other surgical intervention or laser treatment for AMD
Number of eyes treated with brolucizumab | At the brolucizumab index date defined as the date of first brolucizumab injection
  The following types were included:
  OD [eye, right], OS [eye, left], Unspecified, Unilateral, Bilateral)
Number of patient eyes with Visual Acuity (VA) reading | At the brolucizumab index date defined as the date of first brolucizumab injection with lookback of 365 days
  The following categories were included:
  * Snellen: 20/10, 20/12-20/20, 20/25-20/40, 20/50-20/160, ≤20/200
  * Approximate ETDRS letters
Number of patient eyes with Anti-VEGF treatment-naive vs prior-treated | 36-month period prior to the index date (inclusive of the index date) ( index date defined as the date of first brolucizumab injection)
  Anti-VEGF treatment-naive vs prior-treated were measured at the eye level
Number of patient eyes with the prior treatment status | 36-month period prior to the index date (inclusive of the index date) ( index date defined as the date of first brolucizumab injection)
  The following types were included:
  off-label bevacizumab, ranibizumab, aflibercept, unknown, treatment-naive
Number of different prior anti-VEGF agents | 36-month period prior to the index date (inclusive of the index date) ( index date defined as the date of first brolucizumab injection)
  The following categories were measured at the eye level:
  0, 1, 2, ≥3
Number of prior anti-VEGF injections | 36-month period prior to the index date (inclusive of the index date) ( index date defined as the date of first brolucizumab injection)
  Total, per anti-VEGF agent were measured at the eye level)
  * Continuous
  * Categorical: <6, 6 to <12, 12 to <24, ≥24
Duration of last anti-VEGF treatment | 36-month period prior to the index date (inclusive of the index date) ( index date defined as the date of first brolucizumab injection)
  Total, per anti-VEGF agent; will be measured at the eye level
  * All anti-VEGFs i. Continuous ii. Categorical: <6, 6 to <12, 12 to <24, ≥24 months
  * Specific anti-VEGF iii. Continuous iv. Categorical: <6, 6 to <12, 12 to <24, ≥24 months
Time since wet Age-related macular degeneration (AMD) diagnosis | 36-month period prior to the index date (inclusive of the index date) ( index date defined as the date of first brolucizumab injection)
  Patients were measured at the eye level
Time since any Age-related macular degeneration (AMD) diagnosis | 36-month period prior to the index date (inclusive of the index date) ( index date defined as the date of first brolucizumab injection)
  Patients were measured at the eye level
Time from last anti-VEGF injection to index date (among switchers) | At the brolucizumab index date defined as the date of first brolucizumab injection
  The following categories were measured:
  * Continuous (days)
  * Categorical (0-30, 31-60, 61-90, 91+ days)
Number of ocular adverse events (AEs) | Post-index period defined as the 180 days following therapy initiation, excluding index date
  To assess the incidence of ocular AEs among patients treated with brolucizumab

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Pharmaceuticals, East Hanover, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Results for CRTH258AUS15 from the Novartis Clinical Trials Website — http://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17868